### STATISTICAL ANALYSIS PLAN

# "MULTICENTRIC CLINICAL INVESTIGATION ON THE USE OF SINGLE-DOSE OPHTHALMIC SOLUTION BASED ON SODIUM HYALURONATE IN THE TREATMENT OF EYE DISCOMFORT IN PARTICULAR IN CASE OF OCULAR DRYNESS"

Version 1 –October 10<sup>th</sup>, 2023

STUDY CODE: 052/SI Hyalistil Bio PF Mono

Post Market Clinical Follow up (PMCF)

(Observational Study-Profit)

#### **Sponsor**

SIFI SpA Via Ercole Patti 36 95025 Aci S. Antonio (CT) – (Italy) Dr. Fabrizio Chines

**Contract Research Organization** 

Consorzio Universitario Unifarm in Liquidazione

Viale Andrea Doria 21 95125 Catania (Italy) Dr. Santo Ranno

Email: direzione@unifarm.org

Study code: 052/SI Hyalistil Bio PF Mono

| Statistical Analysis Plan Status: DRAFT | |
|---|---|
| Clinical Investigation Plan No.: 052/SI Hyalistil Bi | o PF Mono |
| Study Type: Post Market Clinical Follow up (PMCF) (<br>interventional clinical investigation) | Prospective, observational, non- |
| Products Name: Hyalistil Bio PF Mono | |
| Date of Issue: October 10 <sup>th</sup> , 2023 | |
| Study Title Multicentric clinical investigation on the use of sing sodium hyaluronate in the treatment of eye discomfor Author: | le-dose ophthalmic solution based on<br>7 in particular in case of ocular dryness |
| Statistician, Consorzio Universitario Unifarm in Liquida Name and Surname FILIPPO PALERMO | zione |
| Signature F. L. Fole | Date 10/10/2023 |
| Approval: | The state of the s |
| Scientific Director, Consorzio Universitario Unifarm in I | Liquidazione |
| Name and Surname AGATA KATIA GIUFFRIDA | |
| Signature Agolo Mahio & | Date 13 / 10 / 7073 |
| Approval: | |
| Sponsor Representative, SIFI S.p.A. | |
| Name and Surname GIULIA FARACI | |
| Signature Gulo Foroc' | Date 13 110 12023 |
| Name and Surname LAURA BONINO Signature | Date 13/011/2023 |

# TABLE OF CONTENET

| LIST OF ABBREVIATION | 5 |
|----------------------------------------------------|----|
| 1. CHANGE HISTORY RECORD | 6 |
| 1.1. Statistical Analysis Plan | |
| 1.2. Clinical Investigation Plan | |
| 1.3. CRF | |
| 2. RATIONAL AND BACKGROUND | |
| 3. CLINICAL INVESTIGATION OBJECTIVES | |
| 3.1. Primary objective | |
| 3.2. Secondary objective | |
| 3.3. Safety Evaluations | |
| 4. CLINICAL INVESTIGATION DESIGN | |
| 4.1. Study visits and procedures | |
| 4.2. Treatment Administration | |
| 4.3. Randomization and Blinding | |
| 4.4. Clinical Investigation Scheme | |
| 5. PRIMARY AND SECONDARY OUTCOMES^ | 14 |
| 5.1. Primary Endpoints <sup>#</sup> | 14 |
| 5.2. Secondary Endpoints | 14 |
| 5.3. Safety Endpoints | 15 |
| 6. PLANNED ANALYSIS | 16 |
| 6.1. Interim Analysis | 16 |
| 6.2. Final Analysis | |
| 7. SAMPLE SIZE AND STATISTICAL POWER CONSIDERATION | 16 |
| 8. ANALYSIS POPULATIONS | 16 |
| 8.1. Screening Failures | 16 |
| 8.2 Total Set | 16 |
| 8.3. Intent-to-Treat Population (ITT) | 17 |
| 8.4. Per-Protocol (PP) Population | 17 |
| 8.5. Safety Population | 17 |
| 9. GENERAL ISSUES FOR STATISTICAL ANALYSIS | 17 |
| 9.1 Definitions, Derived Variables and Datasets | 17 |
| 10. STATISTICAL METHODS | |
| 10.1. General Issues for Statistical Analysis | 19 |
| 10.2 Definitions, Derived Variables and Datasets | 19 |
| 10.2.1 Baseline Values | 19 |
| 10.2.2 Demographic Data | 20 |
| 10.2.3 Duration of Exposure | 20 |
| 10.2.4 Treatment Compliance | 20 |
| 10.2.5 . Methods for Withdrawals and Missing Data | 20 |
| 10.2.6. Adverse Events | 20 |
| 10.2.7. Premature Discontinuation | 21 |
| 10.3 Multicenter Studies Considerations | 21 |
| 10.4 Multiple Comparisons and Multiplicity | 21 |
| 10.5 Data Safety Monitoring Board (DSMB) | |
| 11 STUDY PATIENTS | |
| 11.1 Disposition of Patients | 21 |
| 11.2 Protocol Deviations | |
| 12 PERFORMANCE ANALYSIS | 22 |

## Study code: 052/SI Hyalistil Bio PF Mono

| 12.1 | Analysis datasets | |
|----------|-------------------------------------------|----|
| | Demographics and Baseline Characteristics | |
| | Measurements of Treatment Compliance | |
| 13 AN | ALYSIS OF PERFORMANCE | 23 |
| 13.1 | Primary Performance endpoint | 23 |
| 13.2 | Secondary objective | 23 |
| 14. CHA | NGES IN THE PLANNED ANALYSES | 27 |
| 15. LIST | AND SAMPLES OF TABLES, FIGURES AND GRAPHS | 27 |
| 16. LI | ST OF LISTING | 30 |
| 17 REFE | ERENCES | 97 |

Study code: 052/SI Hyalistil Bio PF Mono

## LIST OF ABBREVIATION

| AE Adverse Events CI Confidence intervals DED Dry eye disease DEQS Questionnaire about Eye Symptoms and Daily Life FAS Full Analysis Set IGAS Investigator Global Assessment of Safety IOP Intraocular Pressure ITT Intent-to-Treat LLT Lowest level term LOCF Last observation carried forward method | |
|---|---|
| DED Dry eye disease DEQS Questionnaire about Eye Symptoms and Daily Life FAS Full Analysis Set IGAS Investigator Global Assessment of Safety IOP Intraocular Pressure ITT Intent-to-Treat LLT Lowest level term | |
| DEQS Questionnaire about Eye Symptoms and Daily Life FAS Full Analysis Set IGAS Investigator Global Assessment of Safety IOP Intraocular Pressure ITT Intent-to-Treat LLT Lowest level term | |
| FAS Full Analysis Set IGAS Investigator Global Assessment of Safety IOP Intraocular Pressure ITT Intent-to-Treat LLT Lowest level term | |
| IGAS Investigator Global Assessment of Safety IOP Intraocular Pressure ITT Intent-to-Treat LLT Lowest level term | |
| IOP Intraocular Pressure ITT Intent-to-Treat LLT Lowest level term | |
| ITT Intent-to-Treat LLT Lowest level term | |
| LLT Lowest level term | |
| LOCF Last observation carried forward method | |
| MedDRA Medical Dictionary for Regulatory Activities | |
| NEI National Eye Institute Scale | |
| PP Per Protocol | |
| PPS Per Protocol Set | |
| PT Preferred Term | |
| QOL Quality of Life | |
| SANDE Questionnaire Symptom Assessment in Dry Eye | |
| SAP Statistical Analysis Plan | |
| SEAE Study-emergent adverse event | |
| SD Standard Deviation | |
| SOC System/Organ class | |
| TFBUT Tear Film Break-up Time | ĺ |

## 1. CHANGE HISTORY RECORD

# 1.1. Statistical Analysis Plan

| Statisitcal<br>Analysis<br>Plan<br>version | Statisitcal<br>Analysis<br>Plan<br>date | Description of changes | Amendment version | Amendment<br>date |
|---|---|---|---|---|
| 1 | October 10 <sup>th</sup> 2023 | First version | - | - |

# 1.2. Clinical Investigation Plan

| Clinical<br>Investigation<br>Plan<br>version | Clinical<br>Investigation<br>Plan<br>date | Description of changes | Amendment<br>version | Amendment<br>date |
|---|---|---|---|---|
| 1 | October 10 <sup>th</sup> 2022 | First release | - | - |
| 2 | March 14 <sup>th</sup> ,2023 | Second release | 052/SI Hyalistil Bio PF Mono/EM version 1 of March 14 <sup>th</sup> ,2023 | March 14 <sup>th</sup> ,2023 |

## 1.3. CRF

| CRF<br>version | CRF<br>date | Description of changes | Amendment version | Amendment date |
|---|---|---|---|---|
| 1.0 | March 9 <sup>rd</sup> 2023 | First release | - | - |
| 2.0 | May 29 <sup>th</sup> , 2023 | Second release | | |
| 3.0 | July 24 <sup>th</sup> , 2023 | Third release | | |

#### 2. RATIONAL AND BACKGROUND

Dry eye disease (DED) is a common clinical problem as over 7 million people in the United States experience dry eye symptoms. Symptoms of DED include a sensation of dry eyes, foreign body sensation, irritation, burning, tearing, ocular pain, and itching, among others. DED affects quality of life and work productivity, and patients with moderate to severe DED may experience reduced visual function in addition to ocular dysfunction.

DED is a multi-factorial disease, defined by a loss of homeostasis of the tear film and accompanied by ocular symptoms, in which tear film instability and hyper-osmolarity, ocular surface inflammation and damage, and neuro-sensory abnormalities play etiological roles.

Hyalistil BIO PF (listed in the Medical Device Technical File as HA MONO 0.2% Phosp. Free-) is sterile medical devices (eye drops) for ophthalmic use containing 0.2% sodium hyaluronate. The device is presented in unidose containers phosphate-free. Therefore, HA MONO 0.2% Phosp. Free- is indicated to lubricate and hydrate the ocular surface able to provide a stable coating on the surface of the eye performing a moisturizing and lubricating action on the ocular surface, thus allowing a temporary relief to burning, irritation and all dry-eye related discomfort.

In addition, the device assures the protection of the ocular surface during the healing processes. Moreover, since the presence of phosphates in ophthalmic formulations may rarely cause, in patients with compromised cornea, corneal deposits or corneal opacities [1,2], HA MONO 0.2% Phosp. Free- is a specific formulation without phosphates (and alternative buffer systems) mainly indicated in all cases of ocular discomfort and ocular dryness due to (as example) dry eye syndrome, ocular surgery, allergy, environmental factors (sun exposure, wind, smoke, pollution, conditioned air), excessive use of computer monitors, contact lenses use, aging, Moreover, they protect the ocular surface during the process of wound healing after corneal abrasions.

One-two drops of HA MONO 0.2% Phosp. Free- should be instilled in the conjunctival fornix three to four times daily, unless otherwise indicated.

No safety concerns have been identified and reported on the leaflet with the exception of occasional burning and local irritation upon instillation.

Under these premises, considering that HA-MONO-0.2%-Phosp.free was marketed in Italy with the name "Hyalistil Bio PF", the purpose of this prospective observational investigational plan is to assess the clinical performance, tolerance, and safety of Hyalistil Bio PF device after 35  $\pm$  4 days of treatment in patients affected by eye *discomfort* in particular in case of ocular dryness.

#### 3. CLINICAL INVESTIGATION OBJECTIVES

## 3.1. Primary objective

• Evaluation of Tear film break-up time with fluorescein (TFBUT) at Study Termination Visit ( $Day 35 \pm 4 \text{ of treatment}$ ) compared to Visit 1 (Day 0 of treatment - baseline).

## 3.2. Secondary objective

The secondary objectives were:

#### **Clinical Performance**

- Evaluation of the change in total score (score from 6 to 33, considering a normal score 0-33) resulting from the sum of the corneal staining score (score from 0 to 15) and conjunctival staining score (score from 0 to 18) with fluorescein using the National Eye Institute Scale (NEI) at Visit 2 (Day 14 ± 2 of treatment) and at the Study Termination Visit (Day 35 ± 4 of treatment) compared to Visit 1 (Day 0 of treatment baseline);
- Evaluation of the tear film stability per group as objectified by the tear break up time with fluorescein (TFBUT) at Study Termination Visit (Day  $35 \pm 4$  of treatment) compared to Visit 2 (Day  $14 \pm 2$  of treatment).
- Changes about Best Corrected Visual Acuity (BCVA) measured by the "Early Treatment Diabetic Retinopathy Study" (ETDRS) at Visit 2 (Day 14 ± 2 of treatment) and Study Termination Visit (Day 35 ± 4 of treatment) compared to Visit 1(Day 0 of treatment baseline).

#### **Patient reported outcomes**

- To compare patients reported outcomes (PRO) measures per group, including:
  - Patient's reported symptoms (SANDE) at Visit 2 (*Day 14 ± 2 of treatment*) and Study Termination Visit (*Day 35 ± 4 of treatment*) compared to Visit 1(*Day 0 of treatment baseline*).
  - Evaluation of the degree of satisfaction to the treatment reported by patients through the use of the visual analogue scale (VAS)##, at the Study Termination Visit (*Day 35* ± 4 of treatment).
  - Assessment of the quality of life (QOL)\*\*\*\* by "Questionnaire about Eye Symptoms and Daily Life" (DEQS) at Study Termination Visit (Day  $35 \pm 4$  of treatment) compared to Visit 1 (Day 0 of treatment baseline).

#### 3.3. Safety Evaluations

- Evaluation of safety of daily instillation of ophthalmic solution during all the study period through:
  - ✓ Investigator Global Assessment of Safety (IGAS): using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAS was evaluated at the Study Termination Visit. [Time Frame: Study Termination Visit];
  - ✓ Evaluation of reported adverse events/incidents. [Time Frame: During the treatment period];
  - ✓ Evaluation of intraocular pressure (IOP) [Time frame: Visit 1, Visit 2 and Study

#### Termination Visit];

According to clinical practice, the Investigator will perform all clinical evaluations on both eyes of the individual patient.

In the case that both eyes are affected by ocular dry eye, the statistical analysis will be performed considering the eye with the lowest level of TFBUT score "worse eye". If the level of TFBUT score at baseline is the same in both eyes, then the eye with the highest level of NEI score will be designated as the "worse eye". If the level of NEI score at baseline is the same in both eyes, then the right eye will be designated as the "worse eye."

#### 4. CLINICAL INVESTIGATION DESIGN

This clinical investigation is a multicentric prospective observational open-label, non-interventional clinical investigation evaluation, during the conventional clinical practice, the performance and safety of the daily instillation of Hyalistil Bio PF device in the treatment of patients affected by eye *discomfort* in particular in case of ocular dryness.

The clinical evaluation period was run approximately for 4 months from first patient first visit (FPFV) March 14<sup>th</sup>, 2023, to last patient last visit (LPLV) August 3<sup>tr</sup>, 2023. All patients were followed from enrolment until study end date, which was occur when, in compliance with the normal clinical practice, the last patient was undergo the Study Termination Visit (35± 4 days from the first instillation of study product).

## 4.1. Study visits and procedures

In this observational clinical investigation, each enrolled patient will be evaluated during 3 scheduled visits. A written informed consent will be obtained before any study assessment or procedure. The first patient first visit (FPFV) is defined as the 1st visit to the clinical site by the 1st screened patient. The "Last Patient Last Visit" (LPLV) is defined as the last visit to the clinical site by the last patient (i.e., the last visit foreseen by the study clinical investigation plan), independently of whether the patient completed or withdrew from the study.

#### **Visit 1 (screening-enrolment)**

The following procedures were performed:

- Explanation to the patient of study aims, procedures and possible risks of the observational study;
- Informed consent signature;
- Allocation screening number;
- Demographic data collection;
- In case of female patients (collection of information on pregnancy or breastfeeding self-reported by the patient);
- Medical and surgical history/current medical conditions;
- Prior/concomitant ocular and systemic medications;
- Ocular examination of both eyes:
  - External Ocular Examination;
  - o BCVA test through the ETDRS at 4 m distance;
- o Symptom Assessment in Dry Eye by SANDE questionnaire;

- o Evaluation of Intraocular pressure (IOP);
- o Tear film break-up time with fluorescein (TFBUT)<sup>⋄</sup>;
- o Ocular surface staining (NEI score) with fluorescein;
- DEQS questionnaire administration;
  - Patient eligibility: inclusion/exclusion criteria evaluation;
  - Assignment of the study and allocation patient clinical investigational number;
  - Generation of unique subject identifiers code<sup>-</sup>;
  - Medical device dispensation;
  - Beginning of the treatment\*.

The Investigator will be dispensed to the patients 5 boxes of medical device each containing 30 single-dose containers of medical device for the following 35±4 days. After completing the baseline evaluation, patients will start the study treatment as instructed through self-instillation of medical device under investigation at home\*.

Patients were return to the clinical site on day 14±2 from the first instillation of medical device under investigation (Visit 2).

# Visit 2 (on the 14<sup>th</sup> day from the first instillation of medical device under investigation (MD)) (window $\pm$ 2 days)\*\*\*

The following procedures will be performed:

- Assessment of treatment compliance;
- Current medical conditions;
- Concomitant medications:
- Evaluation of any reported adverse events/incidents\*\*;
- Ocular examination of both eyes:
  - o External Ocular Examination;
  - o BCVA test through the ETDRS at 4 m distance;
  - Symptom Assessment in Dry Eye by SANDE questionnaire;
  - Evaluation of Intraocular pressure (IOP);
  - o Tear film break-up time with fluorescein (TFBUT)<sup>⋄</sup>;
  - Ocular surface staining (NEI score) with fluorescein;

Patients were return to the clinical site on day 35±4 days from the first instillation of medical device under investigation (Study Termination Visit).

# Study Termination Visit (on the $35^{th}$ day from the first instillation of medical device under investigation) (window $\pm 4$ days)

The final visit is defined as the visit performed on  $35 \pm 4$  days after the first instillation of medical device under investigation°.

# <u>In case of premature study discontinuation, patients will undergo an Early Termination Visit (ETV)'.</u>

The following procedures will be performed:

- Assessment of treatment compliance (reconciliation of the amount of used single dose containers and empty/unused medical device boxes returned by patients to the centre)<sup>§</sup>;
- Current medical conditions:

- Concomitant medications:
- Evaluation of any reported adverse events/incidents\*\*;
- Ocular examination of both eyes:
  - o External Ocular Examination;
  - o BCVA test through the ETDRS at 4 m distance;
  - Symptom Assessment in Dry Eye by SANDE questionnaire;
  - o Evaluation of Intraocular pressure (IOP);
  - Tear film break-up time with fluorescein (TFBUT)<sup>6</sup>;
  - o Ocular surface staining (NEI score) with fluorescein;
- Administration of the VAS scale on the degree of satisfaction to the treatment;
- DEQS questionnaire administration;
- Evaluation of the safety of the experimental product through the compilation of the IGAS scale;
- Restitution of remaining medical devices §.
- \* Start of the treatment (window + 1 day).
- \*\* In case of adverse events/incidents all assessments considered necessary by the Investigator was performed, including the possible suspension of treatment.
- \*\*\* Variable because it is based on the planned visit schedule according to clinical practice for the individual patient Visit 2 (windows of  $\pm$  2 days).
- $^{\circ}$  All patients enrolled were treated for 35 days. The Study Termination Visit is variable because it is based on the planned visit schedule according to clinical practice for the individual patient (window  $\pm$  4 days).
- § Restitution of the amount of used single dose containers and empty/unused medical device boxes returned by patients to the centre.

'In case of premature study discontinuation, patients were undergoing an Early Termination Visit (ETV). During the ETV the patients will return the amount of used single dose containers and empty/unused medical device boxes returned by patients to the centre

□ The "unique subject identifiers code" consists of the 5-digit screening number (e.g. S1001, S1002,....S1028 etc.), and, if applicable, the 4-digit subject clinical investigational number (e.g. 1001, 1002,...1028 etc.). Specifically, the first subject clinical investigational number was referred to the study site.

Allocation screening number and subject clinical investigational number are separated by slashes (e.g. "S1001/1001"). (e.g. "S1001/1001" for site number 1, "S2001/2001" for site number 2).

#### 4.2. Treatment Administration

All patients meeting the inclusion and exclusion criteria

### 4.3. Randomization and Blinding

Not applicable: open-label clinical investigation

<sup>&</sup>lt;sup>†</sup> The TFBUT value will be recorded as the average of 3 measurements.

4.4. Clinical Investigation Scheme

| Study Procedure | Visit 1<br>(screening-<br>enrolment- start of<br>treatment)* | Visit 2*** (on the 14 <sup>th</sup> day from the first instillation of medical device) (window ± 2 days) | Study termination Visit° (on the 35 <sup>th</sup> day from the first instillation of medical device) (window ± 4 days) |
|---|---|---|---|
| Informed Consent | $\sqrt{}$ | | |
| Allocation screening number | √ | | |
| Demographic data collection | V | | |
| Medical and surgical history | √ | | |
| Current medical conditions | √ | V | V |
| Prior ocular local and systemic medication | √ | | |
| Concomitant ocular local and systemic medication | | <b>√</b> | √ |
| External Ocular Examination | √ | V | $\sqrt{}$ |
| BCVA evaluation through ETDRS grade | √ | V | |
| SANDE questionnaire | √ | V | V |
| Evaluation of Intraocular pressure (IOP) | V | V | V |
| Ocular surface staining<br>(Fluorescein- NEI score) | V | <b>V</b> | √ |
| Tear Film Break-up Time <sup>6</sup> | V | V | $\sqrt{}$ |
| (TFBUT- Fluorescein) | , | , | • |
| Administration of DEQS### questionnaire | √ | | $\sqrt{}$ |
| Inclusion/Exclusion Criteria | $\sqrt{}$ | | |

Study code: 052/SI Hyalistil Bio PF Mono

| Enrolment and allocation subject clinical | V | | |
|---|---|---|---|
| investigational number | | | |
| Generation of unique subject identifiers | | | |
| code□ | $\checkmark$ | | |
| Medical device dispensing* | V | | |
| Check Compliance (check proper | | | |
| treatment with medical device, use of | | $\sqrt{}$ | $\sqrt{}$ |
| other medication and medical devices) | | | |
| Medical device restitution§' | | | V |
| <b>Evaluation of satisfaction to the treatment</b> | | | 2 |
| by VAS scale | | | V |
| Evaluation of IGAS | | | √ |
| Adverse events /Incidents** | | V | V |

<sup>\*</sup> Start of the treatment (window + 1 day).

'In case of premature study discontinuation, patients will undergo an Early Termination Visit (ETV). During the ETV the patients will return the amount of used single dose containers and empty/unused medical device boxes returned by patients to the centre-

The "unique subject identifiers code" consists of the 5-digit screening number (e.g. S1001, S1002,....S1028 etc.), and, if applicable, the 4-digit subject clinical investigational number (e.g. 1001, 1002,...1028 etc.). Specifically, the first subject clinical investigational number was referred to the study site.

Allocation screening number and subject clinical investigational number are separated by slashes (e.g. "S1001/1001"). (e.g. "S1001/1001" for site number 1, "S2001/2001" for site number 2).

<sup>\*\*</sup> In case of adverse events/incidents all assessments considered necessary by the Investigator will be performed, including the possible suspension of treatment.

<sup>\*\*\*</sup> Variable because it is based on the planned visit schedule according to clinical practice for the individual patient Visit 2 (windows of ± 2 days).

 $<sup>^{\</sup>circ}$  All patients enrolled will be treated for  $35\pm4$  days. The Study Termination Visit is variable because it is based on the planned visit schedule according to clinical practice for the individual patient (window  $\pm4$  days).

<sup>§</sup> Restitution of the amount of used single dose containers and empty/unused medical device boxes returned by patients to the centre.

<sup>&</sup>lt;sup>6</sup> The TFBUT value will be recorded as the average of 3 measurements.

<sup>###</sup>In the event that, for both trial centers, the DEQS questionnaire is not available, the assessment of the quality of the life will be performed by the DEQ-5 questionnaire.

#### 5. PRIMARY AND SECONDARY OUTCOMES^

## 5.1. Primary Endpoints#

• Clinical performance:

-25 % increase from Visit 1 (*Day 0 of treatment - baseline*) to Study Termination Visit (*Day 35*  $\pm$  4 of treatment) of tear film break-up time with fluorescein (TFBUT)  $^{\phi}$  [Time frame: Visit 1 and Study Termination Visit].

For more details see paragraph 13 and the list and samples of tables, figures and graphs, reported in paragraph 15.

## 5.2. Secondary Endpoints

• Reduction from baseline (*Visit 1-Day 0 of treatment*) in the corneal and conjunctival fluorescein staining score using the NEI scale.

Fluorescein staining of the ocular surface is assessed as the total sum of the corneal and conjunctival subregions.

- Corneal Fluorescein Staining (NEI score, sum of 5 subregions, maximum score 15. Each subregion will have a maximum score of 3.

(0=no staining, 3 = maximum staining).

- Conjunctival Fluorescein Staining (NEI score, sum of 6 subregions, maximum score 18. Each subregion will have a maximum score of 3.

(0=no staining, 3 = maximum staining).

[Time frame: Visit 1, Visit 2 and Study Termination Visit].

- Tear film break-up time with fluorescein (TFBUT)<sup>\$\psi\$</sup>. [Time frame: Visit 2 and Study Termination Visit].
- BCVA is measured using the standard Early Treatment Diabetic Retinopathy Study (ETDRS) acuity chart and reported in ETDRS letters. [Time frame: Visit 1, Visit 2 and Study Termination Visit];
- Patient reported outcomes:

Change in intensity## and frequency of dry eye symptoms assessed by completing the questionnaire SANDE. [Time frame: Visit 1, Visit 2 and Study Termination Visit].

- ##In the questionnaire SANDE, the term "intensity" has the same meaning than "severity".
- ###Evaluation of the degree of satisfaction to the treatment reported by patients through the use of the visual analogue scale (VAS) ###, ranging from 0 to 100 mm, at Study Termination Visit (Day  $35 \pm 4$  of treatment). [Time frame: Study Termination Visit].

Patients will be asked to rate their degree of satisfaction to the treatment and answer the following questions:

- "I feel satisfied using this treatment?",
- "With this treatment, I have a feeling of freshness?",
- "With this treatment, I have a feeling of relief?",

#### Study code: 052/SI Hyalistil Bio PF Mono

- "This treatment contributed to reduce my pain due to eye dryness?",
- "This treatment is comfortable?",

Patients will be asked to place a vertical mark on a horizontal line, from 0 to 100 mm, to indicate the degree of satisfaction to the treatment, where:

- $\sqrt{0-10}$  mm=none
- ✓ 11-30 mm=very mild
- ✓ 31-50 mm=mild
- ✓ 51-70 mm=moderate
- $\checkmark$  71-90 mm=strong
- $\checkmark$  91-100 mm=very strong.
- Assessment of the quality of life (QOL) by "Questionnaire about Eye Symptoms and Daily Life" (DEQS) at Study Termination Visit (Day  $35 \pm 4$  of treatment) compared to Visit 1 (Day 0 of treatment baseline). [Time frame: Visit 1 and Study Termination Visit].

For more details see paragraph 13 and the list and samples of tables, figures and graphs, reported in paragraph 15.

###In the event that, for both trial centers, the DEQS questionnaire is not available, the assessment of the quality of the life will be performed by the DEQ 5 questionnaire.

According to clinical practice, the Investigator will perform all clinical evaluations on both eyes of the individual patient.

In the case that both eyes are affected by ocular dry eye, the statistical analysis will be performed considering the eye with the lowest level of TFBUT score "worse eye". If the level of TFBUT score at baseline is the same in both eyes, then the eye with the highest level of NEI score will be designated as the "worse eye". If the level of NEI score at baseline is the same in both eyes, then the right eye will be designated as the "worse eye."

## **5.3.** Safety Endpoints

#### Evaluation of safety parameters

Evaluation of safety of daily instillation of ophthalmic solution during all the study period through:

- Evaluation of safety of daily instillation of ophthalmic solution during all the study period through:
- Investigator Global Assessment of Safety (IGAS): using the 4-point scale:1= very good safety, 2 =good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated at the Study Termination Visit. [Time Frame: Study Termination Visit];
- Evaluation of reported adverse events/incidents. [Time Frame: During the treatment period].
- Evaluation of intraocular pressure (IOP) [Time frame: Visit 1, Visit 2 and Study Termination Visit];
- Evaluation of compliance through verification of correct instillation of the medical device,

#### Study code: 052/SI Hyalistil Bio PF Mono

counting of single dose containers and boxes. [Time Frame: Visit 2 and Study Termination Visit].

^According to clinical practice, the Investigator will perform all clinical evaluations on both eyes of the individual patient.

The statistical analysis will be performed considering right eye as the "study eye."

\*The primary end point will be evaluated on the ITT population and in PP population.

<sup>♦</sup>The TFBUT value will be recorded as the average of 3 measurements.

#### 6. PLANNED ANALYSIS

### **6.1. Interim Analysis**

No interim analysis is planned.

## 6.2. Final Analysis

Final analysis will be performed according to the current version of the protocol (version 2 of March 14<sup>th</sup>, 2023) and to this Statistical Analysis Plan (version 1 of October 10<sup>th</sup>, 2023), after data cleaning operations and Data Base (DB) Lock will be performed.

The statistical analysis will be performed using SAS 9.4 for Windows (SAS Institute Inc., Cary, NC, USA).

#### 7. SAMPLE SIZE AND STATISTICAL POWER CONSIDERATION

A previous study reported by De-Hita-Cantalejo C, et al 2022 [3], baseline level of TFBUT of  $6.23\pm1.75$  in patients with moderate dry eye disease. After 30 days of treatment with tear eyedrops containing hyaluronic acid 0.3%, TFBUT was  $8.10\pm2.06$  s. To detect a 25% of increase of TFBUT at Study Termination Visit compared to the baseline (Visit 1) (mean difference 1.56, s.d. 1,91), considering an alpha = 0.01 (two-tailed) and a power of  $1-\beta=0.80$ , 23 patients are required (Wilcoxon signed-rank test). Taking into account an expected dropout of 20%, it is expected to enroll a total of 28 patients.

#### 8. ANALYSIS POPULATIONS

## 8.1. Screening Failures

Screening failures will be defined as patients who provided informed consent but who were not enrolled randomised. Screening Failures will be summarised and presented by a total count.

More details regarding the patient distribution well be described in the consort figure as reported in paragraph 15.1.

#### 8.2 Total Set

The total set will be defined as all patients who provided informed consent as documented on the 'Informed Consent' eCRF page. The total set will be summarized and presented by a total count (without study treatment categorization).

## 8.3. Intent-to-Treat Population (ITT)

The performance analysis will be performed on the full intent to treat population (ITT) population. The ITT population consisted of all enrolled patients who receive at least one dose of the study experimental product. The patients with no treatment applied at all and the patients who do not have any available data after the first dose of treatment should be excluded from the analysis.

## 8.4. Per-Protocol (PP) Population

The per protocol set (PPS) will be used for supportive performance analysis. The PPS consisted of patients in the ITT who did not have any major protocol violation.

## **8.5.** Safety Population

The safety population, used for all safety analyses, consisted of all patients who received at least one dose of the medical device.

## 9.GENERAL ISSUES FOR STATISTICAL ANALYSIS

#### 9.1 Definitions, Derived Variables and Datasets

| Variable (CRF) | Variable | Type | Description |
|---|---|---|---|
| md_dispensing_q7; checkcomp_and_mdret_q3. | Treat_time | Continuous | Treatment duration |
| age | Age | Continuous | Age |
| sex_at_birth | Sex | Discrete | Sex |
| race | Race | Discrete | Race |
| eoe_q3; eoe_q4; | Ext_oc_ex | Discrete | External ocular examination |
| mh_part1_q1; mh_part1_q1_ongoing; mh_part1_q2; mh_part1_q2_ongoing; mh_part1_q3; mh_part1_q3_ongoing; mh_part1_q4; mh_part1_q4_ongoing; mh_part1_q5; mh_part1_q5; mh_part1_q6; mh_part1_q6; mh_part1_q6_ongoing; otherprevious_cdiseases; table_otherprevious_cd1. | Med_hist | Discrete | Medical history |
| concomitant_q1;<br>concomitant_q2;<br>concomitant_q3; | Conc_med | Discrete | Concomitant medications |

## Study code: 052/SI Hyalistil Bio PF Mono

| concomitant_q4. | | | |
|---|---|---|---|
| tfbut_q2_od; tfbut_q3_od;<br>tfbut_q4_od;<br>tfbut_q2_os; tfbut_q3_os;<br>tfbut_q4_os; | TFBUT | Continuous | Tear film break-up time with fluorescein |
| tfbut_q5_od_a;<br>tfbut_q5_os_a. | | | |
| cornea_od_totalscore_a; cornea_os_totalscore_a; conjunctiva_od_totalscore_c; conjunctiva_od_totalscore_d; cornea_conjunctiva_os_b_d; cornea_conjunctiva_od_a_c; | NEI_total<br>NEI_cornea<br>NEI_conjunt | Continuous | National Eye Institute<br>Scale |
| eoe_q5; | BCVA | Continuous | Best Corrected Visual<br>Acuity |
| sande_q3_severity;<br>sande_q4_frequency;<br>sande_qc_score2; | SANDE_total SANDE_sev SANDE_freq | Continuous | Symptom Assessment in<br>Dry Eye |
| vasscale_q2; vasscale_cornea_q1; vasscale_cornea_q2; vasscale_cornea_q3; vasscale_cornea_q4; vasscale_cornea_q5; | VAS1<br>VAS2<br>VAS3<br>VAS4<br>VAS5 | Continuous | Degree of satisfaction to the treatment |
| sensazione_deqs; secchezzaoculare; doloreagliocchi; stanchezzaoculare; pesantezzadellepalpedre; rossoreagliocchi; sensazione_deqs_1; secchezzaoculare_1; doloreagliocchi_1; stanchezzaoculare_1; rossoreagliocchi_1; deqs_q13; deqs_q14; deqs_q15; deqs_3. GES | DEQS_sum_score<br>DEQS_subscale1<br>DEQS_subscale2 | Continuous | Questionnaire about Eye<br>Symptoms and Daily Life |
| igas_q1 | IGAS | Discrete | (Investigator Global<br>Assessment of Safety) |

Study code: 052/SI Hyalistil Bio PF Mono

| Incident_adverseevent_q1;<br>incident_adverseevents_q2;<br>incident_adverseevent_q3;<br>endofstudy2_q4; | Adv_event_Inc | Discrete | Adverse events/incidents |
|---|---|---|---|
| iop_q2_od; Iop_q2_os; | IOP | Continuous | Evaluation of intraocular pressure |
| checkcompliance_q1;<br>checkcompliance_q2;<br>checkcompl_and_mdret_q3; | Compliance | Continuous/Discrete | Evaluation of compliance through verification of correct instillation of the medical device |

#### 10. STATISTICAL METHODS

Descriptive analysis will be performed by using absolute rate, percentage and frequency tables for qualitative variables.

Normally distributed continuous data will be reported as minimum, maximum, mean and standard deviation, whereas non- normally distributed data as medians and IQR.

Categorical variables will be analyzed by using Yates-corrected chi-square test or Fisher's exact test when appropriate. The McNemar's test will be used to analyze paired nominal data. Differences in endpoints between baseline and different timepoints will be assessed using paired t-test for normally distributed data, whereas the Wilcoxon signed-rank test will be used for non-normally distributed data.

Data distribution will be evaluated through the Kolmogorov-Smirnov test.

A p-value <0.05 will be considered statistically significant.

Analysis will be performed using SAS version 9.4 for Windows (SAS Institute Inc., Cary, NC, USA).

#### 10.1. General Issues for Statistical Analysis

All data will be summarized and listed as appropriate. <del>Performance data will be summarized and listed for the overall population.</del>

Performance data will be summarized, listed and described in table for the overall population.

There are no subgroups.

For more details see paragraph 13 and the list and samples of tables, figures and graphs, reported in paragraph 15.

## 10.2 Definitions, Derived Variables and Datasets

#### 10.2.1 Baseline Values

#### Study code: 052/SI Hyalistil Bio PF Mono

Data collected at the screening/baseline visit (Visit 1), before the beginning of the treatment, are considered as baseline values.

The last observation carried forward method (LOCF) was used to replace missing data in each performance endpoints.

Baseline and demographic characteristics of the patients will be summarized by using appropriate descriptive statistics.

For more details see paragraph 11.1.

## 10.2.2 Demographic Data

Demographic data (age, sex, race) were summarized using mean, SD, minimum, maximum, median, lower quartile and upper quartile for continuous variables and number of patients (frequency) and percentage per category for categorical variables.

## 10.2.3 Duration of Exposure

All patients will be followed from enrolment until study end date, which will occur when, in compliance with the normal clinical practice, the last patient will be patient to the study termination visit (30 days from the first application of study product) (window  $\pm 4$  day).

For each patient enrolled, the duration of exposure per patient will be estimated as the number of days between the first and last treatment administration. Mean and SD, minimum and maximum number of days of treatment will be reported.

## **10.2.4** Treatment Compliance

Treatment duration per patient will be estimated as the number of days between the first and last treatment administration. Absolute rate and percentage of days of treatment will be reported.

Compliance will be estimated as the percentage of administrations given with respect to the administrations planned. Compliance will be also reported categorical as <50%, 50-80% and >80%. In particular:

- 1. < 50% = Poor Compliance
- 2. 50-80% = Moderate Compliance
- 3. > 80% = Good Compliance

Details by patients about compliance well be reported

### 10.2.5. Methods for Withdrawals and Missing Data

Reasons for withdrawal will be considered and patients will be entered in the analysis on the basis the reason for withdrawal.

If the primary performance measurement at Visit 2 is missing, it will be imputed with the score at baseline. If the primary performance measurement at Study Termination Visit is missing, it will be imputed with the score at Visit 2, if it is not missing, or otherwise with the score at baseline.

#### 10.2.6. Adverse Events

Adverse events will be mapped to a Medical Dictionary for Regulatory Activities (MedDRA)

Study code: 052/SI Hyalistil Bio PF Mono

version 19.1 preferred term and system organ classification.

If a patient has multiple adverse events within the same system organ class in the treatment period, the subject will only be counted once at the system organ class level in adverse event frequency tables. Should an event have a missing severity or relationship, it will be classified as having the highest severity and/or strongest relationship to study medication. Summaries of incidence rates (frequencies and percentages) of individual AEs by MedDRA system organ class and preferred term will be prepared. Such summaries will be displayed for all TEAEs, TEAEs by maximum severity, and TEAEs by strongest relationship to clinical investigation medical device.

Serious AEs and AEs leading to discontinuation of investigational product will also be summarized.

All adverse events reported will be listed for individual patients showing both verbatim and preferred terms.

Any adverse event with a missing onset date will be considered to be a TEAE occurring during the treatment period.

#### 10.2.7. Premature Discontinuation

Dropout patients will be defined as patients who prematurely discontinued the study. Patients who had stopped the study treatment but were still being followed in the study were not considered as dropouts.

All data available until the premature discontinuation will be taken into account.

#### 10.3 Multicenter Studies Considerations

Not applicable.

## 10.4 Multiple Comparisons and Multiplicity

When necessary, the multiplicity-adjusted p-value will be calculated by multiplying the unadjusted p-value by the number of times compared.

#### 10.5 Data Safety Monitoring Board (DSMB)

Not applicable.

#### 11 STUDY PATIENTS

#### 11.1 Disposition of Patients

Patient disposition will be presented in terms of the numbers and percentages of patients who completed the study and discontinued from the study patients who are not discontinued from the study will be considered study completers. The disposition of the patients will be described in the

#### CONSORT figure.

The number and percentage of patients prematurely discontinued from the study and the reasons for study discontinuation will be for all enrolled patients. The reasons for study discontinuation that will be summarized include: AE, protocol violation, administrative reasons (e.g., inability to continue, lost to follow up), Sponsor termination of study, patient choice, and other. A patient listing will be provided that includes the date of and reason for premature study discontinuation.

#### 11.2 Protocol Deviations

Protocol deviations will be registered in the monitoring visits reports, performed during the study. Protocol deviations will be described in Table and in Listing.

The number and percentage of patients with any, major, and minor protocol deviations will be summarized for all enrolled patients. Major protocol deviations are defined as protocol deviations that may impact primary performance endpoint; other protocol deviations are classified as minor. Protocol deviations will be assessed prior to database lock and unmasking. The number and percentage of patients with any protocol deviation will also be summarized for the following categories: Informed Consent, Inclusion / Exclusion, Instillation of investigational product. Improper Protocol Procedures at Site, Site's Failure to Report Serious Adverse Event (SAE) / AE, Visit Out of Window, patient's Use of Prohibited Concomitant Medication, and Other. A patient listing will be provided that includes the date, description of each deviation and the classification of whether the deviation was judged to be major or minor.

The Sponsor will consider the following criteria for exclusion of a patient from the PPS:

- Impossibility to assess the compliance with investigational medical product application (patients who have not returned the amount of used single dose containers and/or empty/unused medical device boxes);
- Missing primary performance data;
- Failure to satisfy any inclusion/exclusion criteria;
- Intake of prohibited medications.

#### 12PERFORMANCE ANALYSIS

#### 12.1 Analysis datasets

See Section 10.

#### 12.2 Demographics and Baseline Characteristics

Demographic (age, gender, ethnic origin) and baseline characteristics (vital signs, weight, height, medical history, and physical examination) will be summarized by using minimum, maximum, mean, standard deviation or median and IQR for continuous variables and number of patients and percentage per category for categorical variables.

## **12.3 Measurements of Treatment Compliance**

Details by patients will be reported and compliance will be estimated as the percentage of administrations given with respect to the administrations planned.

Study code: 052/SI Hyalistil Bio PF Mono

Compliance  $(\%) = \frac{Numbers\ of\ vial\ dispensed-Number\ of\ unused\ vials\ returned}{Number\ of\ doses\ planned}$ 

Compliance will be presented categorical as <50% 50-80% and >80%, were:

- 1) <50% = Poor Compliance
- 2) 50-80% = Moderate Compliance
- 3) > 80% = Good Compliance

No further analyses will be planned on compliance. All other collected data including diary information on treatment compliance will be evaluated during the BDRM for relevant protocol deviations and will be listed.

#### 13 ANALYSIS OF PERFORMANCE

## 13.1 Primary performance endpoint

The primary endpoint consists in the assessment of 25 % increase from Visit 1 (*Day 0 of treatment - baseline*) to Study Termination Visit (*Day 35*  $\pm$  4 of treatment) of tear film break-up time with fluorescein (TFBUT). The data will be reported (change vs baseline) as minimum, maximum, mean, standard deviation or median and IQR. According to the data distribution, paired t-test or Wilcoxon signed-rank test will be used to test the statistical significance of the change from baseline to each time points. [Time frame: Visit 1, and Study Termination Visit].

Patients with a Tear Film Break-up Time TFBUT test  $\leq 10$  in the study eye (study eye) at the screening visits are eligible for enrollment.

TFBUT will be measured by determining the time to tear break-up. The TFBUT will be performed after instillation of 5  $\mu$ l of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient will be instructed to blink several times to thoroughly mix the fluorescein with the tear film. To achieve maximum fluorescence, the examiner should wait approximately 30 seconds after instillation before evaluating TFBUT. With the aid of a slit lamp at 10X magnification using cobalt blue illumination, the examiner will monitor the integrity of the tear film, noting the time it takes to form lacunae (clear spaces in the tear film) from the time that the eye is opened after the last blink. This measurement will be performed within 10 seconds maximum. The TFBUT will be measured twice during the first minute after the instillation of the fluorescein. The TFBUT value will be the average of 3 measurements.

#### 13.2 Secondary objective

The secondary objectives were: Clinical Performance

• Changes in NEI score from baseline will be summarized as minimum, maximum, mean,

#### Study code: 052/SI Hyalistil Bio PF Mono

standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank test will be used to test the statistical significance of the change from baseline to each timepoints. [Time frame: Visit 1, Visit 2 and Study Termination Visit].

The cornea is divided into five sectors (central, superior, inferior, nasal and temporal), each of which is scored on a scale of 0–3, with a maximal score of 15. Both nasally and temporally, the conjunctiva is divided into a superior paralimbal area, an inferior paralimbal area and a peripheral area with a grading scale of 0–3 and with a maximal total score of 18 for the nasal and temporal conjunctiva.

For a better reading it is also essential not to use an intense illumination beam, which may reduce the contrast and lead to an underestimation of grading.

- Changes in TFBUT from baseline will be reported as minimum, maximum, mean standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank will be used to test the statistical significance of the change from baseline to each timepoints. [Time frame: Visit 2, and Study Termination Visit].
- Change in the BVCA scores will be summarized as minimum, maximum, mean, standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank test will be used to test the statistical significance. Details of changes (i.e., difference in BVCA scores between baseline and end of treatment) will be summarized as well. [Time frame: Visit 1, Visit 2 and Study Termination Visit].
- Best Corrected Visual Acuity BCVA was measured using the standard Early Treatment Diabetic Retinopathy Study (ETDRS) acuity chart lighting, and procedures and reported in Best-corrected visual acuity is measured at all trial visits using standard charts, (chart 1 is used for testing the visual acuity of the RIGHT eye; Chart 2 for testing the LEFT eye). Patients should not be allowed to see any of the charts before the examination.

A distance of 4 meters is required between the patient's eyes and the visual acuity chart. With the box light off, not more than 15 foot-candles of light (161.4 Lux) should fall on the center of the chart. To measure the amount of light, the room is set up for visual acuity testing, but with the box light off. The light meter is placed at the fourth line from the top of the chart, with its back against the chart and the reading is taken. If more than one line available for testing visual acuity, the visual acuity of an individual patient should be measured in the same line at each visit, if possible. If different lines are used to test visual acuity, they must each meet the same standards.

#### Patient reported outcomes:

• Change in the SANDE scores will be summarized as minimum, maximum, mean, standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank test will be used to test the statistical significance. Details of changes (i.e., difference in SANDE scores between

#### Study code: 052/SI Hyalistil Bio PF Mono

baseline and end of treatment) will be summarized as well. [Time frame: Visit 1, Visit 2 and Study Termination Visit].

The SANDE questionnaire is a short questionnaire to evaluate both the intensity and frequency of dry eye using a 100 mm VAS. The patient's symptoms of ocular dryness and/or irritation will be quantified on the scale based on two questions assessing both severity and frequency of symptoms. For the assessment, patients mark the point that they feel represents their perception of their current state on the 100 mm VAS line. The VAS score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks. The SANDE scores will be then evaluated for the 2 questions severity (0-100) and frequency (0-100). To simplify the procedure the patient will be informed that to provided anchors for the question measuring the frequency of symptoms, the extreme left of the 100 mm line indicated "rarely" and the extreme right indicated "all of the time". Similarly, for the question that measured the severity of symptoms, the words "very mild" and "very severe" were placed at the left and right ends of the 100 mm line, respectively.

At each visit, only one assessment is performed aggregating the situation for both eyes (i.e. no separate assessment per study eye).

Data collected from the SANDE questionnaire were calculated by multiplying the frequency score by the severity score and obtaining the square root.

• VAS will be summarized reporting the number of patients and related percentage in each category. [Time frame: Study Termination Visit].

Patients will be asked to rate their degree of satisfaction to the treatment and answer the following questions:

- "I feel satisfied using this treatment?",
- "With this treatment, I have a feeling of freshness?",
- "With this treatment, I have a feeling of relief?",
- "This treatment contributed to reduce my pain due to eye dryness?",
- "This treatment is comfortable?",

Patients will be asked to place a vertical mark on a horizontal line, from 0 to 100 mm, to indicate the degree of satisfaction to the treatment, where:

- $\sqrt{0-10}$  mm=none
- ✓ 11-30 mm=very mild
- ✓ 31-50 mm=mild
- $\sqrt{51-70}$  mm=moderate
- $\checkmark$  71-90 mm=strong
- $\checkmark$  91-100 mm=very strong.
- Changes from baseline in DEQS for each subscale and total score will be summarized as minimum, maximum, mean, standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank test will be used to test the statistical significance of the change from baseline to the study termination. [Time frame: Visit 1 and Study Termination Visit].

#### Study code: 052/SI Hyalistil Bio PF Mono

The DEQS questionnaire consists of 15 questions divided in two subscales: the Bothersome Ocular Symptoms (six questions) and the Impact on Daily Life (nine questions). Each question is assessed using two-step scales. The first step is to assess the frequency of symptoms and disability, and the second is to assess the degree of severity. The frequency is scored on a 5-point Likert scale ranging from 0 to 4 (0 = never, 4=always). When the answer was "never," then the respondent could skip to the next question; but when any frequency was reported (1–4), the respondent had to rate the degree of severity, which was scored on a 4-point Likert scale ranging from 1 to 4, with a larger number indicating a greater burden.

The total score of the answer will be calculated using the summation of the degree scores of all questions answered multiplied by 25 and divided by the total number of questions answered. The total score ranging from 0 to 100, with a higher score, represented greater disability.

$$Total \ summary \ score = \frac{(Sum \ of \ the \ degree \ scores \ for \ all \ questions \ answeredX \ 25)}{Total \ number \ of \ questions \ answered}$$

Subscale scores will be calculated similarly, using only the item from each subscale.

• GENERAL EYES STATUS (GES) will be summarized as minimum, maximum, mean, standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank test will be used to test the statistical significance of the change from baseline to the study termination. [Time frame: Visit 1 and Study Termination Visit].

GENERAL EYES STATUS will be assessed using the degree scores of a question answered.

GENERAL EYES STATUS will be assessed using the degree scores of a question answered using the 6-point scale: 1= Estremamente bene, 2 = Molto bene, 3 = Bene, 4 = Male, 5= Molto male and 6= Estremamente male.

Safety Evaluation:

- IGAS will be summarized reporting the number of patients and related percentage in each category. [Time frame: Study Termination Visit].

  The Safety of medical device will be assessed using the Investigator Global Assessment of
  - Safety (IGAS): using the 4-point scale:1= very good safety, 2 =good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated during the Study Termination Visit. [Time Frame: Study Termination Visit].
  - Incidents will be coded using the last updated version of the MedDRA dictionary to give a preferred term (PT) and a system/organ class term (SOC) for each event. The number of patients who experienced at least one incident, study product-related incidents, serious incidents, and the number of patients withdrawn due to an incident will be summarized. The frequency of incidents will be presented overall, by SOC and PT, and additional grouping by severity and relationship to the observed treatment will be performed. [Time Frame: During the treatment period].

• Changes from baseline in IOP will be summarized as minimum, maximum, mean, standard deviation or median and IQR. Paired t-test or Wilcoxon signed-rank will be used to test the statistical significance of the change from baseline to each timepoints. [Time frame: Visit 1, Visit 2 and Study Termination Visit].

Intraocular pressure (IOP) measurement was performed using a Goldmann applanation tonometer after topical anesthesia with unpreserved 0.4% oxybuprocaine hydrochloride.

Moreover, for each endpoint, a delta % calculation will be performed.

#### 14. CHANGES IN THE PLANNED ANALYSES

No deviations in the conduct of the study or the planned analysis are anticipated. Should any deviations from the analyses specified in the authorized statistical analysis plan arise, such deviations will be documented in the final clinical study report.

### 15. LIST AND SAMPLES OF TABLES, FIGURES AND GRAPHS

The following lists of tables might not be exhaustive. Additional tables can be produced if necessary.

For each comparison of the various quantitative endpoints (visit 2 versus visit 1 and visit 3 versus visit 1) the descriptive statistics of the endpoint at the two visits will first be calculated and then the P-value will be calculated to assess the statistical significance of the difference. This difference will also be reported as a percentage from baseline.

# 15.1 LIST AND SAMPLES OF FIGURES 1 DISPOSITION OF PATIENTS

Figure 1 Patient's disposition by CONSORT.

#### 15.2 LIST AND SAMPLES OF TABLES

#### 1 TREATMENT DURATION

**Table 1 Treatment duration ITT population** 

#### 2 DEMOGRAPHICS AND OTHER BASELINE DATA

- Table 2.1.1
   Demographic characteristics (screened patients) Age
- Table 2.1.2 Demographic characteristics of Age
- Table 2.1.2 Demographic characteristics (screened patients) Sex
- Table 2.1.3 Demographic characteristics (screened patients) Race
- Table 2.2.1 Demographic characteristics (ITT population) Age
- Table 2.2.2 Demographic characteristics (ITT population) Sex

#### Table 2.2.3 Demographic characteristics (ITT population) Race

- Table 2.3.1 Demographic characteristics (PP population) Age
- Table 2.3.2 Demographic characteristics (PP population) Sex
- Table 2.3.3 Demographic characteristics (PP population) Race
- **Table 2.4.2.1 Medical history (Visit 1: ITT population)**
- Table 2.4.2.2 Medical history (Visit 2: ITT population)
- **Table 2.4.2.3 Medical history (Visit 3: ITT population)**
- **Table 2.4.2.4 Concomitant medications (ITT population)**
- **Table 2.4.3.1 Medical history (Visit 1: PP population)**
- **Table 2.4.3.2 Medical history (Visit 2: PP population)**
- Table 2.4.3.3 Medical history (Visit 3: PP population)
- **Table 2.4.3.4 Concomitant medications (PP population)**

#### 3 COMPLIANCE DATA

- Table 3.1 % Administered doses over the planned doses (ITT population)
- Table 3.2 % Administered doses over the planned doses (PP population)

#### 4 PERFORMANCE DATA (PRIMARY ENDPOINTS)

- Table 4.1.1 TFBUT ITT population (v1) vs (v3)
- Table 4.1.2 Delta % TFBUT ITT population (v1) vs (v3)
- Table 4.2.1 TFBUT PP population (v1) vs (v3)
- Table 4.2.2 Delta % TFBUT PP population (v1) vs (v3)

#### **5 PERFORMANCE DATA (SECONDARY ENDPOINTS)**

- -NEI Scale ITT population
- Table 5.1.1 TOTAL SCORE NEI ITT population (v1) vs (v3)
- Table 5.2.1 TOTAL SCORE NEI ITT population (v1) vs (v2)
- Table 5.3.1 TOTAL SCORE CORNEA ITT population (v1) vs (v3)
- Table 5.3.2 TOTAL SCORE CORNEA ITT population (v1) vs (v2)
- Table 5.4.1 TOTAL SCORE CONJUNCTIVA ITT population (v1) vs (v3)
- Table 5.4.2 TOTAL SCORE CONJUNCTIVA ITT population (v1) vs (v2)

#### -TFBUT ITT POPULATION

Table 5.5.1 TFBUT ITT population (v1) vs (v2)

#### -Questionnaire SANDE ITT population

Table 5.6.1 TOTAL SCORE SANDE ITT population (v1) vs (v3)

Table 5.7.1 TOTAL SCORE SANDE ITT population (v1) vs (v2)

Study code: 052/SI Hyalistil Bio PF Mono

Table 5.8.1 SEVERITY DRYNESS/IRRITATION ITT population (v1) vs (v3) Table 5.8.2 SEVERITY DRYNESS/IRRITATION ITT population (v1) vs (v2)

Table 5.9.1 FREQUENCY DRYNESS/IRRITATION ITT population (v1) vs (v3) Table 5.9.2 FREQUENCY DRYNESS/IRRITATION ITT population (v1) vs (v2)

#### -Questionnaire VAS ITT population

Table 5.10.1 Question "I feel satisfied using this treatment? ", ITT population

Table 5.10.2 Question "With this treatment, I have a feeling of freshness?", ITT population.

Table 5.10.3 Question "With this treatment, I have a feeling of relief?", ITT

Table 5.10.4 Question "This treatment contributed to reduce my pain due to eye dryness?", ITT population

Table 5.10.5 Question "This treatment is comfortable?", ITT population

Table 5.10.6 Total score VAS, ITT population

#### -DEQS ITT POPULATION

Table 5.11.1.1 DEQS Summary score ITT population (v1) vs (v3)

Table 5.11.2.1 DEQS Bothersome Ocular Symptoms subscale ITT population (v1) vs (v3)

Table 5.11.3.1 DEQS Impact on Daily Life subscale ITT population (v1) vs (v3)

Table 5.11.4.1 DEQS-GES ITT population (v1) vs (v3)

#### -IGAS

**Table 5.12.1 IGAS ITT populations** 

#### -IOP ITT POPULATION

Table 5.13.1 IOP ITT population (v1) vs (v3)

Table 5.14.1 IOP ITT population (v1) vs (v2)

Study code: 052/SI Hyalistil Bio PF Mono

## 16. LIST OF LISTING

**Listing 1 ITT Population datasets** 

**Listing 2 PP Population datasets** 

**Listing 3 ITT Population datasets DEQS** 

Listing 4 ITT Population datasets VAS

**FIGURE 1: Patient deposition Screened patients** (n = Screening failures Primary endpoint: (n=0)- Full case (n = xx)- Imputation needed **Included patients (ITT)** (n = xx)Early discontinued (n=xx) (n = xx)Safety set (n = xx)**Excluded** (n = xx)Major protocol deviation (n = xx)**Per Protocol** (n = xx)

Version n.1 dated 10<sup>th</sup> October 2023

Study code: 052/SI Hyalistil Bio PF Mono

Table 1

## ITT population

| Analysis variable: Treatment duration | | | | | | | |
|---|---|---|---|---|---|---|---|
| Mean | Std Dev | Min | Max | N | lower<br>quartile | Median | upper<br>quartile |
| X.XX | X.XX | X.XX | X.XX | XX | X.XX | X.XX | X.XX |
| | | | Test for | <sup>r</sup> Normality | ′ | | |
| 7 | est | | Sta | tistic | P-valu | ue | |
| S | Shapiro-W | ilk | W | x.xxx | Pr < W | X.XXX | |
| k | Kolmogoro | ov-Smirnov | D | x.xxx | Pr > D | x.xxx | |
| ( | Cramer-vo | n Mises | W-Qu | x.xxx | Pr > W-Qu | X.XXX | |
| A | Anderson-l | Darling | A-Qu | X.XXX | Pr > A-Qu | X.XXX | |

Table 2.1.1 Demographics and other baseline data

## **Screened patients**

| Analysis variable: <b>Age</b> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Mean | Std Dev | Min | Max | N | lower<br>quartile | Median | upper<br>quartile |
| X.XX | x.xx | x.xx | x.xx | xx | X.XX | X.XX | X.XX |

| Test for Normality | | | | |
|--------------------|------|-----------|------------|-------|
| Test | | Statistic | P-vai | ue |
| Shapiro-Wilk | W | X.XXX | $Pr \le W$ | x.xxx |
| Kolmogorov-Smirnov | D | x.xxx | Pr > D | x.xxx |
| Cramer-von Mises | W-Qu | x.xxx | Pr > W-Qu | x.xxx |
| Anderson-Darling | A-Qu | x.xxx | Pr > A-Qu | x.xxx |

Table 2.1.2 Demographics and other baseline data

## **Screened patients**

Sex

N %

Male X xx.xx

Female X xx.xx

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

## Table 2.1.3 Demographics and other baseline data

## **Screened patients**

Race

 N
 %

 Caucasian
 x
 xx.xx

 Xxxxx
 x
 xx.xx

 Xxxxx
 x
 xx.xx

Table 2.2.1 Demographics and other baseline data

## **ITT** population

| Analysis variable: <b>Age</b> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Mean | Std<br>Dev | Min | Max | N | lower<br>quartile | Median | upper<br>quartile |
| x.xx | X.XX | x.xx | x.xx | XX | x.xx | x.xx | x.xx |

| Test for Normality | | | | |
|--------------------|------|-----------|------------|-------|
| Test | | Statistic | P-val | ue |
| Shapiro-Wilk | W | x.xxx | $Pr \le W$ | x.xxx |
| Kolmogorov-Smirnov | D | X.XXX | Pr > D | x.xxx |
| Cramer-von Mises | W-Qu | X.XXX | Pr > W-Qu | x.xxx |
| Anderson-Darling | A-Qu | X.XXX | Pr > A-Qu | x.xxx |

## Age (classes, years)

| | Ν | % |
|---------|---|-------|
| [18-64] | Х | xx.xx |
| >65 | Х | xx.xx |

## Age by sex

| | Analysis variable: <b>Age males</b> | | | | | | |
|---|---|---|---|---|---|---|---|
| Mean | Std<br>Dev | Min | Max | N | lower<br>quartile | Median | upper<br>quartile |
| X.XX | X.XX | x.xx | x.xx | XX | x.xx | x.xx | X.XX |

Test for Normality

## Study code: 052/SI Hyalistil Bio PF Mono

| Test | | Statistic | P-vai | lue |
|--------------------|------|-----------|------------|-------|
| Shapiro-Wilk | W | X.XXX | $Pr \le W$ | x.xxx |
| Kolmogorov-Smirnov | D | x.xxx | Pr > D | x.xxx |
| Cramer-von Mises | W-Qu | x.xxx | Pr > W-Qu | x.xxx |
| Anderson-Darling | A-Qu | X.XXX | Pr > A-Qu | X.XXX |

| Analysis variable: <b>Age females</b> | | | | | | | |
|---|---|---|---|---|---|---|---|
| Mean | Std<br>Dev | Min | Max | N | lower<br>quartile | Median | upper<br>quartile |
| x.xx | X.XX | x.xx | x.xx | XX | X.XX | x.xx | X.XX |

| Test for Normality | | | | |
|--------------------|------|-----------|------------|-------|
| Test | | Statistic | P-vai | ue |
| Shapiro-Wilk | W | x.xxx | $Pr \le W$ | x.xxx |
| Kolmogorov-Smirnov | D | x.xxx | Pr > D | x.xxx |
| Cramer-von Mises | W-Qu | x.xxx | Pr > W-Qu | x.xxx |
| Anderson-Darling | A-Qu | x.xxx | Pr > A-Qu | x.xxx |
#### Table 2.2.2 Demographics and other baseline data

## ITT population Sex

Male x xx.xx
Female x xx.xx

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

Table 2.2.3 Demographics and other baseline data

## ITT population Race

 N
 %

 Caucasian
 x
 xx.xx

 xxxxx
 x
 xx.xx

 xxxxx
 x
 xx.xx

Table 2.3.1 Demographics and other baseline data PP population

| | | | | Analysi | is variable: <b>Age</b> | | |
|---|---|---|---|---|---|---|---|
| Mean | Std<br>Dev | Min | Max | N | lower<br>quartile | Median | upper<br>quartile |
| x.xx | x.xx | x.xx | x.xx | XX | x.xx | x.xx | x.xx |

| | Test | for Normalit | y | |
|--------------------|------|--------------|-------------|-------|
| Test | | Statistic | | value |
| Shapiro-Wilk | W | x.xxx | $P_{r} < W$ | X.XXX |
| Kolmogorov-Smirnov | D | x.xxx | Pr > D | x.xxx |
| Cramer-von Mises | W-Qu | x.xxx | Pr > W-Qu | x.xxx |
| Anderson-Darling | A-Qu | x.xxx | Pr > A-Qu | x.xxx |

### Age (classes, years)

 N
 %

 [18-64]
 X
 XX.XX

 >65
 X
 XX.XX

Table 2.3.2 Demographics and other baseline data

Study code: 052/SI Hyalistil Bio PF Mono

## PP population Sex

N %

Male x xx.xx

Female x xx.xx

### Table 2.3.3 Demographics and other baseline data

## PP population Race

| | N | % |
|-----------|---|-------|
| Caucasian | х | XX.XX |
| XXXXX | Х | XX.XX |
| XXXXX | х | XX.XX |

Table 2.4.2.1 Demographics and other baseline data

## ITT population Medical history (Visit 1)

| | N | % |
|-------|---|-------|
| xxxxx | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | Х | XX.XX |

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

Table 2.4.2.2 Demographics and other baseline data

## ITT population Medical history (Visit 2)

| | N | % |
|-------|---|-------|
| XXXXX | Х | XX.XX |
| XXXXX | Х | XX.XX |
| XXXXX | Х | XX.XX |
| XXXXX | Х | XX.XX |
| XXXXX | Х | XX.XX |
| XXXXX | Х | XX.XX |
| XXXXX | Х | XX.XX |

Table 2.4.2.3 Demographics and other baseline data

## ITT population Medical history (Visit 3)

| | N | % |
|-------|---|-------|
| XXXXX | Х | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

Table 2.4.2.4 Demographics and other baseline data

## ITT population Concomitant medications

| | IV | 70 |
|-------|----|-------|
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |

Table 2.4.3.1 Demographics and other baseline data

## PP population

Medical history (Visit 1)

| | N | % |
|-------|---|-------|
| XXXXX | x | XX.XX |
| XXXXX | x | XX.XX |
| XXXXX | x | XX.XX |
| XXXXX | x | XX.XX |
| XXXXX | x | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

Table 2.4.3.2 Demographics and other baseline data

## PP population Medical history (Visit 2)

| | Ν | % |
|-------|---|-------|
| XXXXX | Х | XX.XX |
| xxxxx | X | XX.XX |
| xxxxx | X | XX.XX |
| xxxxx | X | XX.XX |
| xxxxx | X | XX.XX |
| xxxxx | X | XX.XX |
| xxxxx | X | XX.XX |

Table 2.4.3.3 Demographics and other baseline data

## PP population Medical history (Visit 3)

| | N | % |
|-------|---|-------|
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |

Х

XX.XX

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

XXXXX

Table 2.4.3.4 Demographics and other baseline data

## PP population

#### **Concomitant medications**

| | Ν | % |
|-------|---|-------|
| XXXXX | Х | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | X | XX.XX |
| XXXXX | x | XX.XX |
| XXXXX | x | XX.XX |

Table 3.1 % Administered doses over the planned doses

## ITT population % Administered doses over the planned doses

| | | N | % |
|---------|---------------------|---|-------|
| XXXXX | | X | XX.XX |
| XXXXX | | X | XX.XX |
| XXXXX | | X | XX.XX |
| XXXXX | | X | XX.XX |
| XXXXX | | X | XX.XX |
| XXXXX | | Х | XX.XX |
| XXXXX | | Х | XX.XX |
| <50 % | Poor Compliance | х | xx.xx |
| 50-80 % | Moderate Compliance | X | XX.XX |
| > 80 % | Good Compliance | Х | XX.XX |

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

Table 3.2 % Administered doses over the planned doses

## PP population % Administered doses over the planned doses

| 50-80 % | Moderate Compliance | Х | XX.XX |
|---------|---------------------|---|-------|
| <50 % | Poor Compliance | Х | XX.XX |
| | | N | % |
| **** | | * | ^^.^^ |
| XXXXX | | X | XX.XX |
| XXXXX | | Х | XX.XX |
| XXXXX | | Х | XX.XX |
| XXXXX | | X | XX.XX |
| XXXXX | | Χ | XX.XX |
| XXXXX | | Χ | XX.XX |
| XXXXX | | Х | XX.XX |

Program SAS 9.4 ('Local', X64\_10HOME) date xx XXX xxxx

> 80 % Good Compliance

XX.XX

Table 4.1.1 TFBUT ITT population (v1) vs (v3)

## ITT population TFBUT v1 vs v3

Variable: TFBUT Visit 1

| | • | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shapiro-Wilk | | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | | | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ier-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | rson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | x.xx | x.xx | X.XX | x.xx | x.xx | X.XX |

Variable: TFBUT Visit 3

| Test | | | Sta | tistic | P-value | e | |
|---|---|---|---|---|---|---|---|
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Koln | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cran | ner-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | erson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | | Min | Max | Lower quartile | Median | Upper quartile | |
| X | x x.xx x.xx x | | x.xx | X.XX | X.XX | x.xx | X.XX |

#### Variable: Difference TFBUT Visit 3 - Visit 1

| Basic Statistical Measures | | | | |
|---|---|---|---|---|
| Locatio | on | | Variability | |
| Mean | x.xx | Std dev | I | x.xx |
| Median | x.xx | Varian | ce | x.xx |
| Mode | x.xx | Range | | x.xx |
| | | Interqu | x.xx | |
| | Loca | ation test: | Mu0=0 | |
| Test | S | tatistic | P-vai | lue |
| Student's T | t | x.xxx | Pr > t | x.xxxx |
| sign | M | XX | Pr >= M | x.xxxx |
| Signed ran | k S | x.xxx | x.xxxx | |

Program SAS 9.4 ('Local', X64\_10HOME) date xxXXxxxx

Table 4.1.2 Delta % TFBUT ITT population v1-v3

Analysis variable: Delta % TFBUT v1-v3

Mean Std Dev Min Max N Lower quartile Median Upper quartile

x.xx x.xx x.xx x.xx x.xx xx xx x.xx x.xx x.xx x.xx x.xx

Table 4.2.1 TFBUT PP population (v1) vs (v3)

## PP population TFBUT v1 vs v3

Variable: TFBUT Visit 1

| | • | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | | |
| Kolm | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ner-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | erson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | X.XX | X.XX | x.xx | x.xx |

Variable: TFBUT Visit 3

| | Test for Normal | ty | | |
|---|---|---|---|---|
| Test | Statistic | P-valu | е | |
| Shapiro-Wilk | W x.xxx | x Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D x.xxx | x Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu x.xxx | x Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu x.xxx | x Pr > A-Qu | X.XXXX | |
| N Mean Std dev | Min Ma | x Lower quartile | Median | Upper quartile |

Variable: DifferenceTFBUT Visit 3 - Visit 1

| Basic Statistical Measures | | | | |
|---|---|---|---|---|
| Locatio | n | | Variability | |
| Mean | x.xx | Std dev | I | x.xx |
| Median | x.xx | Varian | ce | x.xx |
| Mode | x.xx | Range | | x.xx |
| | | Interquartile range x.xx | | |
| | Loca | tion test: | Mu0=0 | |
| Test | S | tatistic | P-val | ue |
| Student's T | t | x.xxx | $Pr \ge t $ | x.xxxx |
| sign | M | XX | Pr >= M | x.xxxx |
| Signed rank | ς S | x.xxx | x.xxxx | |

Table 4.2.2 Delta % TFBUT PP population v1-v3

| Analysis variable: Delta % TFBUT v1-v3 | | | | | | | |
|---|---|---|---|---|---|---|---|
| Mean | Std Dev | Min | Max | N | Lower quartile | Median | Upper quartile |
| x.xx | X.XX | x.xx | x.xx | XX | X.XX | x.xx | x.xx |

### Table 5.1.1 TOTAL SCORE NEI ITT population (v1) vs (v3)

## **ITT** population

TOTAL SCORE NEI v1 vs v3

#### Variable TOTAL SCORE NEI Visit 1

| | • | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | er-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | erson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | x.xx |

#### Variable: TOTAL SCORE NEI Visit 3

| | Test for | Normality | | |
|--------------------|----------|-----------|----------------|--------|
| Test | Sta | tistic | P-value | e |
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx |
| N Mean Std dev | Min | Max | Lower quartile | Median |

Study code: 052/SI Hyalistil Bio PF Mono

Variable: Difference TOTAL SCORE NEI Visit 3 – Visit 1

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Locati | ion | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |
| Mode | x.xx | C | |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

### Table 5.2.1 TOTAL SCORE NEI ITT population (v1) vs (v2)

### **ITT** population

TOTAL SCORE NEI v1 vs v2

#### Variable TOTAL SCORE NEI Visit 1

| Test | | | Sta | tistic | P-value | e | |
|---|---|---|---|---|---|---|---|
| Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | | |
| Koln | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ner-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | erson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | X.XX | X.XX | x.xx | X.XX |

#### Variable: TOTAL SCORE NEI Visit 2

| Test | Stat | istic | P-value | | |
|---|---|---|---|---|---|
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Variable: Difference TOTAL SCORE NEI Visit 2 - Visit 1

### Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | | |
|---|---|---|---|---|
| Locatio | on | | Variability | |
| Mean | x.xx | Std dev | 7 | x.xx |
| Median | x.xx | Varian | Variance | |
| Mode | x.xx | Range | x.xx | |
| | Interquartile range | | | |
| | Loca | ation test: | Mu0=0 | |
| Test | S | tatistic | P-val | lue |
| Student's T | t | x.xxx | Pr > t | x.xxxx |
| sign | M | $M \qquad xx Pr >= M x$ | | |
| Signed ran | k S | x.xxx | Pr >= S | x.xxxx |

### Table 5.3.1 TOTAL SCORE CORNEA ITT population (v1) vs (v3)

### **ITT** population

TOTAL SCORE CORNEA v1 vs v3

#### Variable TOTAL SCORE CORNEA Visit 1

| Test for Normality | | | | | | |
|---|---|---|---|---|---|---|
| Test | | Sta | tistic | P-value | • | |
| Shapiro-Wilk | | W | x.xxxx | $P_r < W$ | x.xxxx | |
| Kolmogorov-Sm | irnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mise | es | W-Qu | x.xxxx | Pr > W-Qu | X.XXXX | |
| Anderson-Darlin | g | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean St | td dev | Min | Max | Lower quartile | Median | Upper quartile |
| x x.xx | X.XX | x.xx | x.xx | X.XX | x.xx | X.XX |

#### Variable: TOTAL SCORE CORNEA Visit 3

| Test | Stat | istic | P-value | | |
|---|---|---|---|---|---|
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Variable: Difference TOTAL SCORE CORNEA Visit 3 – Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| | Basic Statistical Measures | | |
|---|---|---|---|
| Locati | ion | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | X.XX |
| Location test: Mu0=0 | | | |

Test Statistic P-value

Student's T t x.xxx Pr > |t| x.xxxx

 $sign \hspace{1cm} M \hspace{1cm} xx \hspace{1cm} Pr >= |M| \hspace{1cm} x.xxxx$ 

Signed rank  $S = x.xxx = Pr \ge |S| = x.xxxx$ 

### Table 5.3.2 TOTAL SCORE CORNEA ITT population (v1) vs (v2)

### **ITT** population

TOTAL SCORE CORNEA v1 vs v2

#### Variable TOTAL SCORE NEI Visit 1

| Test for Normality | | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | • | |
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ier-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | X.XX | X.XX | x.xx | x.xx |

#### Variable: TOTAL SCORE CORNEA Visit 2

| Test | Stat | tistic | P-value | | |
|---|---|---|---|---|---|
| Shapiro-Wilk | W | X.XXXX | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Variable: Difference TOTAL SCORE CORNEA Visit 2 - Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|---|---|---|---|
| Locati | ion | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |
| - | | | |
| | Location test: Mu0=0 | | |

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr >= |M|x.xxxxSigned rankSx.xxxPr >= |S|x.xxxx

## Table 5.4.1 TOTAL SCORE CONJUNCTIVA ITT population (v1) vs (v3) ITT population

TOTAL SCORE CONJUNCTIVA v1 vs v3

#### Variable TOTAL SCORE CONJUNCTIVA Visit 1

| Test | Statis | tic | P-value | ) | |
|--------------------|--------|-------|----------------|--------|--------------|
| Shapiro-Wilk | W x | x.xxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D x | x.xxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu x | x.xxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu x | x.xxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quarti |
| x x.xx x.xx | X.XX | X.XX | x.xx | X.XX | X.X |

#### Variable: TOTAL SCORE CONJUNCTIVA Visit 3

| Test for Normality | | | | | |
|---|---|---|---|---|---|
| Test | Statistic | | P-value | • | |
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| x x.xx x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |

Study code: 052/SI Hyalistil Bio PF Mono

#### Variable: Difference TOTAL SCORE CONJUNCTIVA Visit 3 - Visit 1

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Locati | ion | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

Test Statistic P-value

Student's T t x.xxx Pr > |t| x.xxxx

Sign  $M \times x \cdot Pr \ge |M| \cdot x.xxxx$ 

Signed rank  $S = x.xxx = Pr \ge |S| = x.xxxx$ 

### Table 5.4.2 TOTAL SCORE CONJUNCTIVA ITT population (v1) vs (v2)

### **ITT** population

TOTAL SCORE CONJUNCTIVA v1 vs v2

#### Variable TOTAL SCORE CONJUNCTIVA Visit 1

| Test for Normality | | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | • | |
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | ogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx |

#### Variable: TOTAL SCORE CONJUNCTIVA Visit 2

| | Test for I | Normality | | | |
|---|---|---|---|---|---|
| Test | Stat | tistic | P-value | • | |
| Shapiro-Wilk | W | X.XXXX | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Variable: Difference TOTAL SCORE CONJUNCTIVA Visit 2 - Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Location | | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

### Table 5.5.1 TFBUT ITT population (v1) vs (v2)

### **ITT** population

TFBUT v1 vs v2

#### Variable TFBUT Visit 1

| Test for Normality | | | | | | | • |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Koln | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ner-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | erson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx | X.XX |

#### Variable: TFBUT Visit 2

| | Test for | Normality | | |
|--------------------|----------|-----------|----------------|--------|
| Test | Sta | tistic | P-value | e |
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx |
| N Mean Std dev | Min | Max | Lower quartile | Median |

Variable: Difference TFBUT Visit 2 – Visit 1

#### Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Locati | ion | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

### Table 5.6.1 TOTAL SCORE SANDE ITT population (v1) vs (v3)

## **ITT** population

TOTAL SCORE SANDE v1 vs v3

#### Variable TOTAL SCORE SANDE Visit 1

| | = | | |
|--------------------|-------------|-----------------------|----------------|
| Test | Statistic | P-value | |
| Shapiro-Wilk | W x.xxxx | Pr < W x.xxxx | |
| Kolmogorov-Smirnov | D x.xxxx | $P_r > D$ x.xxxx | |
| Cramer-von Mises | W-Qu x.xxxx | Pr > W-Qu x.xxxx | |
| Anderson-Darling | A-Qu x.xxxx | Pr > A-Qu $x.xxxx$ | |
| N Mean Std de | v Min Max | Lower quartile Median | Upper quartile |
| x x.xx x.x | x.xx x.xx | x.xx x.xx | X.XX |

#### Variable: TOTAL SCORE SANDE Visit 3

| | Test for I | Normality | | | |
|---|---|---|---|---|---|
| Test | Sta | tistic | P-value | • | |
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Study code: 052/SI Hyalistil Bio PF Mono

Variable: Difference TOTAL SCORE SANDE Visit 3 – Visit 1

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Location Variability | | | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

## Table 5.7.1 TOTAL SCORE SANDE ITT population (v1) vs (v2) ITT population

TOTAL SCORE SANDE v1 vs v2

#### Variable TOTAL SCORE SANDE Visit 1

| | • | | | | |
|---|---|---|---|---|---|
| Test | Sta | atistic | P-value | Э | |
| Shapiro-Wilk | W | x.xxxx | $Pr \le W$ | x.xxxx | |
| Kolmogorov-Smirn | v D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std o | ev Min | Max | Lower quartile | Median | Upper quartile |
| x x.xx x. | x x.xx | x.xx | x.xx | X.XX | X.XX |

#### Variable: TOTAL SCORE SANDE Visit 2

| | • | | | | |
|--------------------|------|--------|----------------|--------|-------------|
| Test | Sta | tistic | P-value | e | |
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quart |
| x x.xx x.xx | x.xx | X.XX | x.xx | X.XX | х.> |

Study code: 052/SI Hyalistil Bio PF Mono

Variable: Difference TOTAL SCORE SANDE Visit 2 - Visit 1

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Locati | on | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

# Table 5.8.1 SEVERITY DRYNESS/IRRITATION ITT population (v1) vs (v3) ITT population

SEVERITY DRYNESS/IRRITATION v1 vs v3

#### Variable SEVERITY DRYNESS/IRRITATION Visit 1

| | Test for Normality | | = |
|---|---|---|---|
| Test | Statistic | P-value | |
| Shapiro-Wilk | W x.xxxx | Pr < W x.xxxx | |
| Kolmogorov-Smirnov | D x.xxxx | Pr > D $x.xxxx$ | |
| Cramer-von Mises | W-Qu x.xxxx | Pr > W-Qu $x.xxxx$ | |
| Anderson-Darling | A-Qu x.xxxx | Pr > A-Qu $x.xxxx$ | |
| N Mean Std dev | Min Max | Lower quartile Median | Upper quarti |
| x x.xx x.xx | x.xx x.xx | x.xx x.xx | X.X |

#### Variable: SEVERITY DRYNESS/IRRITATION Visit 3

| Test | | Statistic | | P-value | | | |
|---|---|---|---|---|---|---|---|
| Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | | |
| Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx |

Study code: 052/SI Hyalistil Bio PF Mono

#### Variable: Difference SEVERITY DRYNESS/IRRITATION Visit 3 – Visit 1

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Locati | ion | Variability | |
| Mean | X.XX | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | X.XX |

Location test: Mu0=0

Test Statistic P-value

Student's T t x.xxx Pr > |t| x.xxxx

Sign  $M \times x \cdot Pr >= |M| \cdot x.xxxx$ 

Signed rank  $S = x.xxx = Pr \ge |S| = x.xxxx$ 

### Table 5.8.2 SEVERITY DRYNESS/IRRITATION ITT population (v1) vs (v2)

### **ITT** population

SEVERITY DRYNESS/IRRITATION v1 vs v2

#### Variable SEVERITY DRYNESS/IRRITATION Visit 1

| | Test for Normality | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | Statistic | | P-value | | | |
| Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | | |
| Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N I | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx |

#### Variable: SEVERITY DRYNESS/IRRITATION Visit 2

| | Test for I | Normality | | | |
|---|---|---|---|---|---|
| Test | Statistic | | P-value | | |
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Variable: Difference SEVERITY DRYNESS/IRRITATION Visit 2 – Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|----------------------------|----|---------------------|------|
| Locati | on | Variability | |
| Mean x.xx | | Std dev | x.xx |
| Median x.xx | | Variance | x.xx |
| Mode x.xx | | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

# Table 5.9.1 FREQUENCY DRYNESS/IRRITATION ITT population (v1) vs (v3) ITT population

FREQUENCY DRYNESS/IRRITATION v1 vs v3

#### Variable FREQUENCY DRYNESS/IRRITATION Visit 1

| Test for Normality | | | |
|---|---|---|---|
| Test | Statistic | P-value | |
| Shapiro-Wilk | W x.xxxx | Pr < W x.xxxx | |
| Kolmogorov-Smirnov | D x.xxxx | Pr > D $x.xxxx$ | |
| Cramer-von Mises | W-Qu x.xxxx | Pr > W-Qu $x.xxxx$ | |
| Anderson-Darling | A-Qu x.xxxx | Pr > A-Qu $x.xxxx$ | |
| N Mean Std dev | Min Max | Lower quartile Median | Upper quarti |
| x x.xx x.xx | x.xx x.xx | x.xx x.xx | X.X |

#### Variable: FREQUENCY DRYNESS/IRRITATION Visit 3

| | | | Test for | Normality | | | |
|---|---|---|---|---|---|---|---|
| Test | | Statistic | | P-value | | | |
| Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | | |
| Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | X.XX | X.XX | X.XX | X.XX |
Study code: 052/SI Hyalistil Bio PF Mono

#### Variable: Difference FREQUENCY DRYNESS/IRRITATION Visit 3 – Visit 1

| 1 | Basic Statistical Measures | | |
|---|---|---|---|
| Location | | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

Test Statistic P-value

Student's T t x.xxx Pr > |t| x.xxxx

Sign  $M \times x \cdot Pr >= |M| \cdot x.xxxx$ 

Signed rank  $S = x.xxx = Pr \ge |S| = x.xxxx$ 

# Table 5.9.2 FREQUENCY DRYNESS/IRRITATION ITT population (v1) vs (v2)

# **ITT** population

FREQUENCY DRYNESS/IRRITATION v1 vs v2

#### Variable FREQUENCY DRYNESS/IRRITATION Visit 1

| Test | | | Sta | tistic | P-value | e | |
|---|---|---|---|---|---|---|---|
| Shapi | ro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | ogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | er-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Ande | rson-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | X.XX | X.XX | x.xx | X.XX |

#### Variable: FREQUENCY DRYNESS/IRRITATION Visit 2

| Test | Statistic | | P-value | | |
|---|---|---|---|---|---|
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |

Variable: Difference FREQUENCY DRYNESS/IRRITATION Visit 2 – Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Locati | ion | Variability | |
| Mean | X.XX | Std dev | x.xx |
| Median | X.XX | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

Table 5.10.1 VAS Question "I feel satisfied using this treatment? ", ITT population

| VAS1 | | |
|-----------------------|---|------|
| | N | % |
| 0-10 mm=none | X | x.xx |
| 11-30 mm=very mild | X | X.XX |
| 31-50 mm=mild | X | x.xx |
| 51-70 mm=moderate | X | x.xx |
| 71-90 mm=strong | X | x.xx |
| 91-100 mm=very strong | X | X.XX |

Program SAS 9.4 ('Local', X64\_10HOME) date xxXXXxxxx

Table 5.10.2 VAS Question "With this treatment, I have a feeling of freshness?", ITT population

| VAS2 | | |
|-----------------------|---|------|
| | Ν | % |
| 0-10 mm=none | x | x.xx |
| 11-30 mm=very mild | X | X.XX |
| 31-50 mm=mild | X | X.XX |
| 51-70 mm=moderate | X | x.xx |
| 71-90 mm=strong | X | X.XX |
| 91-100 mm=very strong | X | X.XX |

Study code: 052/SI Hyalistil Bio PF Mono

Table 5.10.3 VAS Question "With this treatment, I have a feeling of relief?", ITT population

| VAS3 | | |
|-----------------------|---|------|
| | N | % |
| 0-10 mm=none | X | X.XX |
| 11-30 mm=very mild | X | X.XX |
| 31-50 mm=mild | X | x.xx |
| 51-70 mm=moderate | X | X.XX |
| 71-90 mm=strong | X | x.xx |
| 91-100 mm=very strong | X | x.xx |

Table 5.10.4 VAS Question "This treatment contributed to reduce my pain due to eye dryness?"", ITT population

| VAS4 | | |
|-----------------------|---|------|
| | N | % |
| 0-10 mm=none | X | x.xx |
| 11-30 mm=very mild | X | X.XX |
| 31-50 mm=mild | X | x.xx |
| 51-70 mm=moderate | X | X.XX |
| 71-90 mm=strong | X | X.XX |
| 91-100 mm=very strong | X | x.xx |

Program SAS 9.4 ('Local', X64\_10HOME) date xxXXXxxxx

Table 5.10.5 VAS Question "This treatment is comfortable?, ITT population

| VAS5 | | |
|-----------------------|---|------|
| | N | % |
| 0-10 mm=none | X | x.xx |
| 11-30 mm=very mild | X | X.XX |
| 31-50 mm=mild | X | X.XX |
| 51-70 mm=moderate | X | x.xx |
| 71-90 mm=strong | X | x.xx |
| 91-100 mm=very strong | X | x.xx |

Study code: 052/SI Hyalistil Bio PF Mono

Table 5.10.6 Total score VAS, ITT population

| | | tal score VAS | variable: <b>To</b> | Analysis v | | | |
|---|---|---|---|---|---|---|---|
| upper<br>quartile | Median | lower<br>quartile | N | Max | Min | Std Dev | Mean |
| X.XX | X.XX | x.xx | xx | x.xx | X.XX | X.XX | x.xx |

| Test for Normality | | | | |
|--------------------|------|-----------|------------|-------|
| Test | | Statistic | P-val | ue |
| Shapiro-Wilk | W | x.xxx | $Pr \le W$ | x.xxx |
| Kolmogorov-Smirnov | D | x.xxx | Pr > D | x.xxx |
| Cramer-von Mises | W-Qu | x.xxx | Pr > W-Qu | x.xxx |
| Anderson-Darling | A-Qu | x.xxx | Pr > A-Qu | x.xxx |

Table 5.11.1.1 DEQS Summary score ITT population (v1) vs (v3)

# **ITT** population

DEQS Summary score v1 vs v3

### Variable DEQS Summary score Visit 1

| Test | | | Sta | tistic | P-value | e | |
|---|---|---|---|---|---|---|---|
| Shapir | o-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmo | gorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Crame | r-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anders | son-Da | rling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | X.XX | X.XX | x.xx | X.XX |

### Variable: DEQS Summary score Visit 3

| Test for Normality | | | |
|---|---|---|---|
| Test | Statistic | P-value | |
| Shapiro-Wilk | W x.xxxx | Pr < W x.xxxx | |
| Kolmogorov-Smirnov | D x.xxxx | Pr > D $x.xxxx$ | |
| Cramer-von Mises | W-Qu x.xxxx | Pr > W-Qu $x.xxxx$ | |
| Anderson-Darling | A-Qu x.xxxx | Pr > A-Qu $x.xxxx$ | |
| N Mean Std dev | Min Max | Lower quartile Median | Upper quartile |
| x x.xx x.xx | x.xx x.xx | x.xx x.xx | X.XX |
| Shapiro-Wilk Kolmogorov-Smirnov Cramer-von Mises Anderson-Darling N Mean Std dev | W x.xxxx D x.xxxx W-Qu x.xxxx A-Qu x.xxxx | Pr < W x.xxxx $Pr > D$ x.xxxx $Pr > W$ -Qu x.xxxx $Pr > A$ -Qu x.xxxx $Pr > A$ -Qu $Pr > A$ | Upper quartil |

Variable: Difference DEQS Summary score Visit 3 – Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Location | | Variability | |
| Mean | X.XX | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

Table 5.11.2.1 DEQS Bothersome Ocular Symptoms subscale ITT population (v1) vs (v3)

## ITT population

DEQS subscale1 v1 vs v3

#### Variable DEQS subscale1 Visit 1

| | Test for Normality | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shap | Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Koln | Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | x.xx | X.XX | x.xx | x.xx |

#### Variable: DEQS subscale1 Visit 3

| Test | Sta | tistic | P-value | | |
|---|---|---|---|---|---|
| Shapiro-Wilk | W | x.xxxx | Pr < W | x.xxxx | |
| Kolmogorov-Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| x x.xx x.xx | x.xx | X.XX | x.xx | x.xx | x.xx |

Variable: Difference DEQS subscale1 Visit 3 - Visit 1

Study code: 052/SI Hyalistil Bio PF Mono

| Basic Statistical Measures | | | |
|----------------------------|------|---------------------|------|
| Location | | Variability | |
| Mean | X.XX | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valu=Student's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

Table 5.11.3.1 DEQS Impact on Daily Life subscale ITT population (v1) vs (v3)

# **ITT** population

DEQS subscale2 v1 vs v3

#### Variable DEQS subscale2 Visit 1

| Test for Normality | | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | nogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | x.xx | x.xx | X.XX | X.XX | x.xx | X.XX |

### Variable: DEQS subscale2 Visit 3

| | • | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | Statistic P-value | | e | |
| Shap | iro-Wilk | | W | x.xxxx | $P_r < W$ | x.xxxx | |
| Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | x.xx | x.xx | X.XX | x.xx | X.XX | x.xx |

Variable: Difference DEQS subscale2 Visit 3 – Visit 1

### Study code: 052/SI Hyalistil Bio PF Mono

| 1 | Basic Statistical Measures | | |
|--------|----------------------------|---------------------|------|
| Locati | on | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |
| | | _ | |

Location test: Mu0=0

Test Statistic P-value

Student's T t x.xxx Pr > |t| x.xxxx

sign  $M \times x \cdot Pr \ge |M| \cdot x.xxxx$ 

Signed rank  $S = x.xxx = Pr \ge |S| = x.xxxx$ 

# Table 5.11.4.1 DEQS GES ITT population (v1) vs (v3)

# **ITT** population

DEQS GES v1 vs v3

#### Variable DEQS GES Visit 1

| Test for Normality | | | | | |
|---|---|---|---|---|---|
| Test | St | atistic | P-value | e | |
| Shapiro-Wilk | W | x.xxxx | $Pr \le W$ | x.xxxx | |
| Kolmogorov-Smiri | ov D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | |
| N Mean Std | ev Mir | Max | Lower quartile | Median | Upper quartile |
| x x.xx x | XX X.XX | x.xx | x.xx | x.xx | x.xx |

### Variable: DEQS GES Visit 3

| | • | | | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shap | iro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Koln | Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | |
| Cramer-von Mises | | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | x.xx | x.xx | X.XX | x.xx | X.XX | x.xx |

Variable: Difference DEQS GES Visit 3 – Visit 1

### Study code: 052/SI Hyalistil Bio PF Mono

| 1 | Basic Statistical Measures | | |
|----------|----------------------------|---------------------|------|
| Location | | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

 $\begin{tabular}{llll} \textit{Test} & \textit{Statistic} & \textit{P-value} \\ \\ Student's T & t & x.xxx & Pr > |t| & x.xxxx \\ \\ sign & M & xx & Pr > = |M| & x.xxxx \\ \\ \end{tabular}$ 

Signed rank  $S = x.xxx = Pr \ge |S| = x.xxxx$ 

Study code: 052/SI Hyalistil Bio PF Mono

Table 5.12.1 IGAS Investigator Global Assessment of Safety, ITT population

| IGAS | | |
|--------------------|---|------|
| | N | % |
| 1 very good safety | X | x.xx |
| 2 good safety | X | x.xx |
| 3 moderate safety | X | x.xx |
| 4 poor safety | X | X.XX |

# Table 5.13.1 IOP Intraocular Pressure, ITT population (v1) vs (v3)

# **ITT** population

IOP v1 vs v3

#### Variable IOP Visit 1

| | | | Test for | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | | |
| Koln | Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ner-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx |

### Variable: IOP Visit 3

| | | | Test for | | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shap | Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Koln | Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ner-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | x.xx | x.xx | X.XX | X.XX | x.xx | X.XX |

### Study code: 052/SI Hyalistil Bio PF Mono

Variable: Difference IOP Visit 3 - Visit 1

| Basic Statistical Measures | | |
|---|---|---|
| on | Variability | |
| x.xx | Std dev | x.xx |
| x.xx | Variance | x.xx |
| x.xx | Range | x.xx |
| | Interquartile range | x.xx |
| | x.xx<br>x.xx | x.xx Std dev x.xx Variance x.xx Range |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

# Table 5.14.1 IOP Intraocular Pressure, ITT population (v1) vs (v2)

# **ITT** population

IOP v1 vs v2

#### Variable IOP Visit 1

| | | | Test for | Test for Normality | | | |
|---|---|---|---|---|---|---|---|
| Test | Test | | | tistic | P-value | e | |
| Shap | Shapiro-Wilk | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | ogorov- | Smirnov | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | er-von N | Mises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | x.xx | X.XX | x.xx | X.XX | X.XX | x.xx | X.XX |

### Variable: IOP Visit 2

| | | | Test for | Test for Normality | | | |
|---|---|---|---|---|---|---|---|
| Test | | | Sta | tistic | P-value | e | |
| Shapiro-Wilk | | | W | x.xxxx | Pr < W | x.xxxx | |
| Kolm | Kolmogorov-Smirnov | | D | x.xxxx | Pr > D | x.xxxx | |
| Cram | ier-von N | /lises | W-Qu | x.xxxx | Pr > W-Qu | x.xxxx | |
| Anderson-Darling | | A-Qu | x.xxxx | Pr > A-Qu | x.xxxx | | |
| N | Mean | Std dev | Min | Max | Lower quartile | Median | Upper quartile |
| X | X.XX | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx |

### Study code: 052/SI Hyalistil Bio PF Mono

Variable: Difference IOP Visit 2 - Visit 1

| | Basic S | Statistical Measures | |
|--------|---------|----------------------|------|
| Locati | ion | Variability | |
| Mean | x.xx | Std dev | x.xx |
| Median | x.xx | Variance | x.xx |
| Mode | x.xx | Range | x.xx |
| | | Interquartile range | x.xx |

Location test: Mu0=0

TestStatisticP-valueStudent's Ttx.xxxPr > |t|x.xxxxsignMxxPr > = |M|x.xxxxSigned rankSx.xxxPr > = |S|x.xxxx

# Sample listing

Listings will be issued as PDF files. Mock listings are reported in the following section.

| | | | | | | g 1 IT | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | VISIT | VAR 1 | VAR 2 | VAR 3 | VAR 4 | VAR 5 | VAR 6 | VAR 7 | VAR 8 | VAR 9 | VAR<br>10 | VAR<br>11 | VAR<br>12 | VAR<br>13 |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | -xx.x | XX | XX | XX | XX.X | -xx.x |
| XXxxx- | X | XX | XX | XX.X | XX | XX | XX | XX.X | -xx.x | Х | Х | Х | X.X | -xx.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | X.X | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | X | XX | XX | XX.X | XX | XX | XX | xx.x | XX.X | XX | XX | XX | xx.x | -x.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | х.х | XX | XX | XX | xx.x | X.X |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | -x.x | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | X.X | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | X.X | XX | XX | XX | xx.x | -xx.x |
| XXXX- | Х | XX | XXX | XX.X | XX | XX | XX | XX.X | -x.x | XX | XX | XX | xx.x | X.X |
| XXXXX- | Х | XX | XX | XX.X | XX | XX | xx | XX.X | XX.X | XX | XX | XX | xx.x | х.х |
| XXxxx- | X | XX | XX | XX.X | XX | XX | XX | XX.X | -xx.x | XX | XX | XX | XX.X | -xx.x |
| XXxxx- | X | XX | XX | XX.X | XX | XX | XX | XX.X | -xx.x | XX | Х | Х | X.X | -xx.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | -x.x | XX | Х | Х | х.х | -xx.x |

## Study code: 052/SI Hyalistil Bio PF Mono

| | | | | | | | | ulatio | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | VISIT | VAR 1 | VAR 2 | | | | | | | | VAR<br>10 | VAR<br>11 | VAR<br>12 | VAR<br>13 |
| XXxxx-<br>xxx | Х | XX | XX | XX.X | XX | XX | XX | XX.X | -xx.x | XX | XX | XX | XX.X | -xx. |
| XXXX- | Х | XX | XX | xx.x | XX | XX | XX | XX.X | -xx.x | Х | Х | Х | х.х | -xx. |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | X.X | XX | XX | XX | XX.X | -xx. |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | XX.X | XX | XX | XX | XX.X | -x.2 |
| XXXXX- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | x.x | XX | XX | XX | xx.x | х.х |
| XXXXX- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | -x.x | XX | XX | XX | xx.x | -xx. |
| XXXXX- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | x.x | XX | XX | XX | xx.x | -xx. |
| XXXXX- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | x.x | XX | XX | XX | xx.x | -xx. |
| XXXX- | Х | XX | XXX | xx.x | XX | XX | XX | XX.X | -x.x | XX | XX | XX | XX.X | х.х |
| XXXXX- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | xx.x | XX | XX | XX | xx.x | х.х |
| XXXXX- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | -xx.x | XX | XX | XX | xx.x | -xx. |
| XXXX- | Х | XX | XX | xx.x | XX | XX | XX | XX.X | -xx.x | XX | Х | Х | х.х | -xx. |
| XXXX- | Х | XX | XX | xx.x | XX | XX | XX | XX.X | -x.x | XX | Х | Х | X.X | -xx. |

| | | | | | _ | | _ | | ataset | | S | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | VISIT | VAR 1 | VAR 2 | VAR 3 | VAR 4 | VAR 5 | VAR 6 | VAR 7 | VAR 8 | VAR 9 | VAR<br>10 | VAR<br>11 | VAR<br>12 | VAR<br>13 |
| XXxxx-<br>xxx | Х | XX | XX | XX.X | XX | XX | XX | XX.X | -xx.x | XX | XX | XX | XX.X | -xx.x |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | -xx.x | Х | Х | Х | х.х | -xx.x |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | х.х | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | xx.x | XX | XX | XX | xx.x | -x.x |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | X.X | XX | XX | XX | xx.x | х.х |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | -x.x | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | X.X | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | X.X | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | xxx | xx.x | XX | XX | XX | xx.x | -x.x | XX | XX | XX | xx.x | X.X |
| XXxxx- | Х | XX | XX | xx.x | XX | XX | XX | xx.x | XX.X | XX | XX | XX | xx.x | X.X |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | -xx.x | XX | XX | XX | xx.x | -xx.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | xx.x | -xx.x | XX | Х | Х | х.х | -xx.x |
| XXxxx- | Х | XX | XX | XX.X | XX | XX | XX | XX.X | -x.x | XX | Х | Х | X.X | -xx.x |

## Study code: 052/SI Hyalistil Bio PF Mono

| | | | | Populatio | | | | |
|---|---|---|---|---|---|---|---|---|
| PATIENT | VISIT | VAR 1 | VAR 2 | VAR 3 | VAR 4 | VAR 5 | VAR 6 | VAR 7 |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | xx.x |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | xx.x | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | xx.x | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | xx.x | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | xx.x | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XXX | xx.x | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |
| XXxxx-xxx | X | XX | XX | XX.X | XX | XX | XX | XX.X |

Study code: 052/SI Hyalistil Bio PF Mono

### 17 REFERENCES

- 1. Schrage NF, et al Changing the composition of buffered eye-drops prevents undesired side effects. Br J Ophthalmol. 2010; 94:1519-1522,
- 2. EMA/CHMP/753373/2012, Questions and answers on the use of phosphates in eye drops
- 3. De-Hita-Cantalejo C, et al. Performance of hyaluronic acid 0.3%, cyanocobalamin, electrolytes, and P-Plus in menopause patients with moderate dry eye disease. Graefes Arch Clin Exp Ophthalmol. 2022 Feb;260(2):529-535.
- 4. Yuri Sakane, et al. Development and Validation of the Dry Eye–Related Quality-of-Life Score Questionnaire JAMA Ophthalmol. 2013;131(10):1331-1338.